CLINICAL TRIAL: NCT00424853
Title: Randomized Phase II Trial of Two Sequential Schedules of Docetaxel and Cisplatin Followed by Gemcitabine in Patients With Advanced Non-small-cell Lung Cancer.
Brief Title: ADVANCED Phase II Trial of Weekly vs 3 Weekly Docetaxel and Cisplatin Followed by Gemcitabine in Non-small-cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Medical Director, Sanofi-aventis administrative office
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976B_2506; EudraCT # : 2004-001044-72
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

ARMS (2):
- A (Experimental)
  Interventions: Drug: Docetaxel and cisplatin followed by gemcitabine
- B (Experimental)
  Interventions: Drug: docetaxel and cisplatin followed by gemcitabine

INTERVENTIONS:
Drug: Docetaxel and cisplatin followed by gemcitabine — docetaxel 75 mg/m2 day 1 + cisplatin 75 mg/m2 day1 repeated every 21 days for 3 cycles followed by gemcitabine 1200 mg/m2 day 1,8 repeated every 21 days for 3 cycles
  Arms: A
Drug: docetaxel and cisplatin followed by gemcitabine — docetaxel 25 mg/m2 day 1,8,15 + cisplatin 25 mg/m2 days1,8,15 repeated every 28 days for 3 cycles followed by gemcitabine 1200 mg/m2 day 1,8 repeated every 21 days for 3 cycles.
  Arms: B

SUMMARY:
This is a multicenter, open-label, randomized phase II trial whose aim is to assess the antitumor activity of two sequential schedules of docetaxel and cisplatin followed by gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC; Histologic subtypes may include large cell, squamous cell, or adenocarcinoma or a generic cytological diagnosis of NSCLC;
* Patients must have a locoregionally advanced unresectable non metastatic NSCLC Stage IIIB (only N3 supraclavicular or T4 for pleural effusion) or Stage IV according to the revised International Staging System;
* Patients must have at least one measurable lesion according to RECIST criteria.
* Previous radical surgery (more 30 days before study entry) is allowed but a pathologic proof of progression of neoplastic disease must be documented;
* WHO Performance Status 0 or 1 ;
* Weight loss < 5% within the last 3 months;
* Laboratory requirements at entry

  * Blood cell counts: Absolute neutrophils > 2.0 . 10^9/L; Platelets > 100 . 10^9/L; Hemoglobin > 10 g/dl
  * Renal function: Serum creatinine < 1 upper normal limits (UNL). In case of limit value of serum creatinine, the creatinine clearance should be > 60 mL/min
  * Hepatic functions: Serum bilirubin < 1 x UNL; ASAT and ALAT < 2.5 x UNL; Alkaline phosphatase < 5 x UNL (unless accompanied by extensive bone metastases)

Exclusion Criteria:

* Prior systemic chemotherapy or immunotherapy ; prior neoadjuvant or adjuvant chemotherapy is allowed if ended at least 12 months before enrollment;
* Prior radiotherapy for NSCLC to measurable lesions. Prior radiotherapy (to < 25% of the bone marrow) is allowed in non target lesions. At least 4 weeks must be elapsed since the completion of the radiotherapy and the patient must have all side effects recovered.
* Cyto-histological diagnosis of small cell lung cancer, carcinoid, or mixed small-cell / non-small cell lung cancer;
* Patients with evaluable, not measurable disease only (non target lesions);
* Patients with symptomatic brain metastases or with leptomeningeal disease;
* History of prior malignancies, except for cured non melanoma skin cancer, curatively treated in situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least five years;
* History of hypersensitivity reaction to polysorbate 80;
* Pregnant or lactating women (women of childbearing potential must use adequate contraception);
* Current peripheral neuropathy NCI grade > 2;
* Significant neurological or psychiatric disorders ;
* Participation in clinical trials with other experimental agents within 30 days of study entry;
* Other serious concomitant illness of medical conditions:

  1. Uncontrolled cardiovascular disease;
  2. History of significant neurologic or psychiatric disorders including demential or seizures;
  3. Active infection requiring iv antibiotics;
  4. Active ulcer, unstable diabetes mellitus or other contra-indication to corticotherapy;
  5. Any other condition which in the judgement of the investigator would place the subject at undue risk or interfere with the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2005-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
overall response rate assessed by RECIST criteria. | before, during and at the end of treatment

SECONDARY OUTCOMES:
Time to progression | from the date of randomization to the date of first documented tumor progression or relapse
time to treatment failure | from the date of treatment start to the date of diagnosis of progression, withdrawal from study treatment for any reason, administraztion of other antitumor treatment, or death for any cause
overall survival | time interval from the date of randomisation to the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Georges Paizis, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Milan, Italy